CLINICAL TRIAL: NCT02552407
Title: Thrombectomy in ST Elevation Myocardial Infarction, an Individual Patient Meta-analysis
Status: Completed | Type: Observational
Sponsor: Population Health Research Institute (Other)
Collaborators: Uppsala University (Other); Region Örebro County (Other); University Medical Center Groningen (Other); University of Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: ThrombectomyMetaAnalysis
Record Dates: First submitted 2015-09-10; First posted 2015-09-17 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Myocardial Infarction; Acute Coronary Syndromes
Keywords: thrombectomy; acute coronary syndromes; percutaneous coronary intervention; STEMI
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Manual Aspiration Thrombectomy with PCI: Subjects from the randomized controlled trials to be included in this meta-analysis will have been randomly allocated to Manual Aspiration Thrombectomy followed by percutaneous coronary intervention (PCI).
  Interventions: Device: Manual Aspiration Thrombectomy
- PCI Alone: Subjects from the randomized controlled trials to be included in this meta-analysis will have been randomly allocated to percutaneous coronary intervention (PCI) alone without manual aspiration thrombectomy.

INTERVENTIONS:
Device: Manual Aspiration Thrombectomy — Thrombus aspiration
  Groups: Manual Aspiration Thrombectomy with PCI

SUMMARY:
During primary percutaneous coronary intervention, distal embolization of thrombus and impaired microvascular perfusion has been associated with an increased mortality. Thrombectomy devices during primary percutaneous coronary intervention may prevent distal embolization by reducing thrombus burden and thus improve microvascular perfusion and reduce mortality.

DETAILED DESCRIPTION:
An individual patient meta-analysis of large randomized controlled trials comparing manual thrombectomy versus percutaneous coronary intervention alone in patients with ST elevation myocardial infarction will provide significantly more power to detect differences in mortality as well as important but rare events such as stroke and to assess benefits in pre-defined subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Randomized controlled trials comparing manual thrombectomy vs. percutaneous coronary intervention alone in patients with ST elevation myocardial infarction published between January 1980 and April 2015.
* Large trials randomizing more than 1000 patients.
* Trials must have had at least 30 day follow up.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ST elevation myocardial infarction undergoing emergency percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 18000 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Occurrence of Cardiovascular death | up to 30 days
  time to event analysis

SECONDARY OUTCOMES:
Occurrence of Cardiovascular death | up to 180 days
  time to event analysis

OTHER OUTCOMES:
Occurrence of Stroke | up to 30 days
  time to event analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sanjit S Jolly, MD, Principal Investigator — Population Health Research Institute

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jolly SS, James S, Dzavik V, Cairns JA, Mahmoud KD, Zijlstra F, Yusuf S, Olivecrona GK, Renlund H, Gao P, Lagerqvist B, Alazzoni A, Kedev S, Stankovic G, Meeks B, Frobert O. Thrombus Aspiration in ST-Segment-Elevation Myocardial Infarction: An Individual Patient Meta-Analysis: Thrombectomy Trialists Collaboration. Circulation. 2017 Jan 10;135(2):143-152. doi: 10.1161/CIRCULATIONAHA.116.025371. Epub 2016 Dec 9. PMID 27941066